CLINICAL TRIAL: NCT04928898
Title: The First United Arab Emirates National Representative Birth Cohort Study
Acronym: UAE-BCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Ayesha Salem Al Dhaheri, Professor, United Arab Emirates University
Other Study IDs: UAE-BCS
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Child and Maternal Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, a multidisciplinary team of researchers was established including credible researchers from the UAE, Australia and the United Kingdom to launch the First United Arab Emirates 3-year birth cohort study. The study aims to recruit 250 pregnant Emirati women within their first trimester, which is defined by the study as from 8 to 12 weeks pregnant, recruited from obstetric and gynaecology clinics in the UAE. Participants will be recruited via face to face interviews and will receive a total of 11 visits with 1 visit in each trimester of pregnancy and 8 visits after delivery. Maternal data collection includes, socio-demographic and lifestyle factors, dietary intake, anthropometric measurements, physical activity, maternal psychological state, and blood samples for biochemical analysis. Post-partum, visits will take place when the child is 0.5, 4, 6, 9, 12, 18, and 24 months old, with data collection including infant anthropometric measurements, young child feeding practices, dietary intake, supplement use and the eating environment at home, as well as all maternal data collection described above, apart from blood samples. Additional data collection for the child includes developmental assessments taking place at three timepoints, 1) within 2 weeks of birth, 2) at 10-14 months and 3) at 22 - 26 months of age. Developmental assessments for the infant include vision, health, neurological examination, neurodevelopmental and sleep assessments.

ELIGIBILITY:
Inclusion Criteria:

* Emirati Nationality
* Within first trimester of pregnancy (between 8 -12 weeks of gestation)
* Singleton pregnancy
* Absence of major illness preconception (Diabetes mellitus, hypertension, kidney disease, cancer, epilepsy, severe psychiatric illness, and other chronic diseases of infections such as autoimmune disorders, human immunodeficiency virus, and hepatitis).

Exclusion Criteria:

* Non-Emirati
* Unconfirmed viable, intrauterine pregnancy at first obstetric ultrasound during first trimester
* Twin or multiple gestation pregnancy and a history of multiple gestations
* History of chronic illness (i.e., T2DM, hypertension, etc.)
* Previously given birth to babies with malformation, intellectual disability, or inborn errors of metabolism.
* Experience of a miscarriage before 28 weeks of gestation
* On significant regular medications, including insulin, anti-hypertensive agents, psychotropic medications, anti-epileptic drugs, steroids, immune-suppressive agents, and chemotherapeutic agents.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study aims to recruit a total of 250 pregnant Emirati females during their first trimester (8 - 12 weeks of gestation) through face-to-face recruitment at OB-GYN clinics in selected health care facilities across the emirates of the UAE. The participants will be provided with both verbal and written information (Participant Information sheet) about the study aims, data collected, and duration of the study. Mothers will provide written consent on behalf of their children to be included in the study. Participants will give consent by signing the study consent form after their agreement and after meeting the following inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maternal Dietary Intake | 1st Trimester One point during weeks 1 - 13
  24 hour dietary recall
Maternal Dietary Intake | 2nd Trimester. One point during Weeks 14 - 26
  24 hour dietary recall
Maternal Dietary Intake | 3rd Trimester One point during weeks 27 - 42
  24 hour dietary recall
Maternal Dietary Intake | 4 months post natal
  24 hour dietary recall
Maternal Dietary Intake | 18 months post natal
  24 hour dietary recall
Maternal Dietary Intake | 1st Trimester - One point during weeks 1 - 13
  Food frequency questionnaire
Maternal Dietary Intake | 2nd Trimester. One point during Weeks 14 - 26
  Food frequency questionnaire
Maternal Dietary Intake | 3rd Trimester One point during weeks 27 - 42
  Food frequency questionnaire
Maternal Dietary Intake | 4 months post natal
  Food frequency questionnaire
Maternal Dietary Intake | 18 months post natal
  Food frequency questionnaire
Maternal Weight | 1st Trimester - One point during weeks 1 - 13
  Measured in Kilograms
Maternal Weight | 2nd Trimester. One point during Weeks 14 - 26
  Measured in Kilograms
Maternal Weight | 3rd Trimester One point during weeks 27 - 42
  Measured in Kilograms
Maternal Weight | 0.5 months post natal
  Measured in Kilograms
Maternal Weight | 4 months post natal
  Measured in Kilograms
Maternal Weight | 6 months post natal
  Measured in Kilograms
Maternal Weight | 9 months post natal
  Measured in Kilograms
Maternal Weight | 12 months post natal
  Measured in Kilograms
Maternal Weight | 18 months post natal
  Measured in Kilograms
Maternal Weight | 24 months post natal
  Measured in Kilograms
Maternal Blood Pressure | 1st Trimester - One point during weeks 1 - 13
  Measured sphygmomanometer, in millimetres of mercury.
Maternal Blood Pressure | 2nd Trimester. One point during Weeks 14 - 26
  Measured sphygmomanometer, in millimetres of mercury.
Maternal Blood Pressure | 3rd Trimester One point during weeks 27 - 42
  Measured sphygmomanometer, in millimetres of mercury.
Maternal Physical Activity | 2nd Trimester. One point during Weeks 14 - 26
  International Physical Activity Questionnaire
Maternal Physical Activity | 12 months post natal
  International Physical Activity Questionnaire
Maternal Physical Activity | 24 months post natal
  International Physical Activity Questionnaire
Child neurodevelopmental assessment | 24 months post-natal
  INTERGROWTH-21st Neurodevelopment Assessment
Child neurodevelopmental assessment | 12 months post-natal
  Oxford Neonatal Neurodevelopmental Assessment tool
Child neurodevelopmental assessment | 0.5 months post-natal
  Neonatal Neurodevelopmental Assessment tool
Child anthropometric assessment (MUAC) | 0.5 months post-natal
  Weight (kgs), length, head circumference, mid-upper arm circumference
Child anthropometric assessment (MUAC) | 4 months post-natal
  Weight (kgs), length, head circumference, mid-upper arm circumference
Child anthropometric assessment (MUAC) | 6 months post-natal
  Weight (kgs), length, head circumference, mid-upper arm circumference
Child anthropometric assessment (MUAC) | 9 months post-natal
  Weight (kgs), length, head circumference, mid-upper arm circumference
Child anthropometric assessment (MUAC) | 12 months post-natal
  Weight (kgs), length, head circumference, mid-upper arm circumference
Child anthropometric assessment (MUAC) | 18 months post-natal
  Weight (kgs), length, head circumference, mid-upper arm circumference
Child anthropometric assessment (MUAC) | 24 months post-natal
  Weight (kgs), length, head circumference, mid-upper arm circumference

SECONDARY OUTCOMES:
Maternal hemoglobin | 1st Trimester - One point during weeks 1 - 13
  Hemoglobin levels measured in grams per deciliter
Maternal hemoglobin | 3rd Trimester One point during weeks 27 - 42
  Hemoglobin levels measured in grams per deciliter
Maternal Ferritin | 1st Trimester - One point during weeks 1 - 13
  Serum ferritin measured in nanograms per milliliter
Maternal Ferritin | 3rd Trimester One point during weeks 27 - 42
  Serum ferritin measured in nanograms per milliliter
Maternal Folate | 1st Trimester - One point during weeks 1 - 13
  Serum folate measured in nanograms per milliliter
Maternal Folate | 3rd Trimester One point during weeks 27 - 42
  Serum folate measured in nanograms per milliliter
Maternal Vitamin D | 1st Trimester - One point during weeks 1 - 13
  Serum 25 hydroxyvitamin D measured in nanomole per liter
Maternal Vitamin D | 3rd Trimester One point during weeks 27 - 42
  Serum 25 hydroxyvitamin D measured in nanomole per liter
Maternal Vitamin A | 1st Trimester - One point during weeks 1 - 13
  Serum retinol measured in micrograms of retinol activity equivalent
Maternal Vitamin A | 3rd Trimester One point during weeks 27 - 42
  Serum retinol measured in micrograms of retinol activity equivalent
Maternal Vitamin B12 | 1st Trimester - One point during weeks 1 - 13
  Serum B12 measured in picogram per millilitre
Maternal Vitamin B12 | 3rd Trimester One point during weeks 27 - 42
  Serum B12 measured in picogram per millilitre
Maternal zinc concentration | 1st Trimester - One point during weeks 1 - 13
  Serum zinc measured in micromole per litre
Maternal zinc concentration | 3rd Trimester One point during weeks 27 - 42
  Serum zinc measured in micromole per litre
Maternal lead concentration | 3rd Trimester One point during weeks 27 - 42
  Serum lead measured in micromole per litre

CONTACTS AND LOCATIONS:
Locations (1):
- United Arab Emirates University, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No